CLINICAL TRIAL: NCT04660981
Title: The Effect of the Training Program Provided to Primipara Pregnant Women Through the Motivational Interview Method on Their Fear of Childbirth, Childbirth Self-Efficacy and Delivery Mode: A Randomized Controlled Study
Brief Title: The Effect of the Training Program Provided to Primipara Pregnant Women Through the Motivational Interview Method on Their Fear of Childbirth, Childbirth Self-Efficacy and Delivery Mode
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Pelin Calpbinici, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018.05.48
Record Dates: First submitted 2020-11-25; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Fear of Childbirth; Childbirth Self-efficacy; Mode of Delivery; Motivational Interview
MeSH Terms: interventions — Prenatal Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): The women in the intervention group were individually provided with "Training Program on Fear of Childbirth Based on Motivational Interview Method" once a week, four sessions in total.
  Interventions: Behavioral: Antenatal education
- Control Group (No Intervention): No interventions were made for those in the control group other than routine hospital practices.

INTERVENTIONS:
Behavioral: Antenatal education — Training Program on Fear of Childbirth Based on Motivational Interview Method
  Arms: İntervention Group

SUMMARY:
This two-group, parallel randomized controlled study was conducted to evaluate the effect of the training program provided to primipara pregnant women through the motivational interview method on their fear of childbirth, childbirth self-efficacy and delivery mode. The primipara pregnant women included in the study sample were assigned to the intervention (n=37) and control (n=36) groups using the block randomization method. The women in the intervention group were individually provided with "Training Program on Fear of Childbirth Based on Motivational Interview Method" once a week, four sessions in total, while no interventions were made for those in the control group other than routine hospital practices. Study data were collected using a descriptive information form, the Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) versions A-B, the Childbirth Self-Efficacy Inventory-Short Form (CBSEI-SF) and the Delivery Evaluation Form. The value of p<0.05 was accepted statistically significant in the data analyses.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and write in Turkish
* Not contraindicated for vaginal delivery
* Absence of any pregnancy-related complications
* Absence of chronic systemic disease
* Absence of communication problems
* Absence of psychiatric problems
* No abnormalities in the fetus
* 24th and 28th weeks of pregnancy

Exclusion Criteria:

* Premature birth (before 37th weeks of gestation)
* Pregnancy complication developed at any stage of the study (such as preeclampsia, placenta previa, oligohydramnios, gestational diabetes)
* A cesarean section is planned at any stage of the study due to a medical indication,
* Did not complete the training program
* Giving birth outside the province
* Not seen within 24 hours after birth

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 73 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) A version | Change from the WDEQ A scores at pre-training (24th and 28th gestational week), post-training (4 weeks later) and 37th and 40th gestational week
  W-DEQ Version A, which was developed in Sweden in 1998 by Wijma and Klaas, was adapted into Turkish by Körükçü et al. in 2009. It is a 6-point Likert type scale and consists of 33 items. The answers in the scale are scored from 0 to 5, with 0 indicating "completely" and 5 indicating "none." The minimum score on the scale is 0, whereas the maximum score is 165. A high total score indicates a high level of fear; 85 points are considered as the cut-off value. A score of ≥85 indicates clinical level fear.
Childbirth Self-Efficacy Inventory-Short Form (CBSEI-SF) | Change from the CBSEI-SF scores at pre-training (24th and 28th gestational week), post-training (4 weeks later) and 37th and 40th gestational week
  The short form of the Childbirth Self-efficacy Inventory has two subscales: outcome expectancy and efficacy expectancy (Ip, et al., 2008). Efficacy expectancy (EE) is a personal conviction about one's ability to successfully perform the required behaviors in a given situation, and outcome expectancy (OE) is the belief that a given behavior will lead to a given outcome. Each subscale consists of 16 items and yields a score between 16 and 160. Higher scores indicate higher levels of efficacy or outcome efficacy for birth.
The Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ) B version | W-DEQ-B scores at postpartum first day
  The W-DEQ-B was created by Wijma and et al. to evaluate intrapartum childbirth fear in the postpartum period. The validity and reliability study of the scale was conducted by Körükçü et al. It is composed of 32 items. It uses a 6-point Likert scale: 0 corresponds to completely, and 5 corresponds to never. The lowest and the highest scores for the scale are 0 and 160, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans.